CLINICAL TRIAL: NCT00409162
Title: A Prospective, Open Label, Non Randomized, First-In-Man (Feasibility) Study to Evaluate the Safety and Effectiveness of the Eraser Tattoo Removal Device
Brief Title: Safety and Efficacy Study of a New Device for Tattoo Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Hawk Medical Technologies Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA 3722; 91/06; HM-AHR-1 Rev. 02
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Tattoo; Healthy
Keywords: Tattoo removal

INTERVENTIONS:
Device: Eraser TM device, with washing fluid

SUMMARY:
A new mechanical device is evaluated for tattoo removal, comparing two types of needle washing fluids. 30 healthy subjects with tattoos will be treated. The study hypothesis is that the device can be used to achieve satisfactory tattoo removal.

DETAILED DESCRIPTION:
The new device (Eraser TM) uses multiple needles action with a washing fluid to remove tattoos. Healthy patients who wish to remove a tattoo will be enrolled. The study will test the removal of a small part of the tattoo (5cm2 area). Treatment lasts about 20 minutes (with local analgesia if needed), after which an absorptive bandage is put over the treated area for an hour and removed. Treatment may be performed using one of two washing fluids. For one of them, blood samples for material blood level will be taken before and several times after treatment. Pictures of the tattooed area being removed will be taken before and after treatment, and at each follow-up evaluation.

Follow up evaluations will be performed at 1 week, two weeks, one month and two months post treatment. Overall health and skin condition will be evaluated, and the tattoo area will be pictured. Efficacy of tattoo removal will be evaluated after two months, by visual estimation of the percent area that reacted to treatment, and the change in brightness (both evaluated on a 1-5 analog scale). Depending on the result of tattoo removal, and on skin condition, the study treatment will be stopped (if treatment is successful), or may be repeated (up to a limit of two additional times) if the tattoo was not completely removed.

The results of tattoo removal using both washing fluids will be analyzed and compared. A result of 3 or more on the brightness change scale will be considered as a successful treatment.

Pharmacokinetic data for washing fluid no. 2 will be collected and analyzed, to provide Cmax and AUC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older, of any race
* Subject has a tattoo for removal on the back, shoulders or abdomen (areas that can usually be hidden)
* Subjects willing to participate as evidenced by signing the written informed consent

Exclusion Criteria:

* Subject has a dermatological disease, active or latent (e.g. psoriasis)
* Subject has a known tendency for Keloid formation.
* Subject has a known tendency for skin hyperpigmentation.
* Subject is susceptible to Koebner reaction.
* Subject has blood transmittable diseases (HIV, HBV, HCV, etc.)
* Subject has known allergy to device components/ treatment fluids
* Subject has medical conditions that may be worsened by concomitant use of washing fluid, or worsened by local anesthesia materials.
* Subject is taking certain medications or topical preparations.
* Female subject who is pregnant or lactating.
* Subject participating in any other clinical study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-12; Study Completion 2007-10

PRIMARY OUTCOMES:
Pigment clearance, as evaluated by image comparison on a 1-5 analog scale
Rate of systemic and dermatologic adverse events
Pharmacokinetic data for washing fluid (Cmax and AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Shay Efrati, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Research & Development Unit, Assaf-Harofeh Medical Center,, Ẕerifin, Israel